CLINICAL TRIAL: NCT04438317
Title: Thoracic Drains in Intensive Care Units. Comparison of Seldinger and Surgical Methods: A Prospective Randomized Multicenter Study
Brief Title: Thoracic Drains in Intensive Care Units: Comparison of Seldinger and Surgical Methods
Acronym: DrainICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DrainICU - RBHP 2019 GODET 2
Record Dates: First submitted 2020-06-03; First posted 2020-06-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-12

CONDITIONS: Pleural Effusion; Pneumothorax; Hemothorax
Keywords: Pleural effusion; Pneumothorax; Hemothorax; Intensive Care Unit; Seldinger; Drain; Chest drainage; Complications; Comparison of chest drainage techniques in ICU patients; Small drain inserted by Seldinger technique; Large drains inserted by surgical-like technique
MeSH Terms: conditions — Pleural Effusion; Pneumothorax; Hemothorax

STUDY DESIGN:
Intervention Model Description: * Prospective clinical trial, randomized, controlled, open-label
  * Two parallel groups, comparing two strategy involving different medical devices
Who Masked: Outcomes Assessor
Masking Description: Since the study is based on two different techniques, the masking of participants, care providers and local investigator is impossible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seldinger Technique (Active Comparator): Small bore chest tubes inserted by Seldinger technique. A needle is inserted into the intercostal space, and the aspiration of a fluid allows the confirmation the correct position, possibly after ultrasound tracking. A metal guidewire is inserted through the needle, which is then removed. A dilator is then inserted on the metal guidewire to dilate the skin and the subcutaneous tissues. The chest tube is finally inserted on the guide, which is finally removed, and the chest tube is connected to the aspiration system after fixation to the chest wall.
  Interventions: Procedure: Pleural drainage procedure with Seldinger procedure
- Surgical-like Technique (Active Comparator): Large bore chest tube inserted by surgical-like technique. Progressive chest wall dissection is conducted with appropriate instruments (scissors, scalpel, clamps…) by a non-surgeon physician. Large bore drain with rigid introductor is blindly inserted in the pleural cavity, secured to the chest wall with suture fixation and further connection to the aspiration system.
  Interventions: Procedure: Pleural drainage procedure with surgical-like technique

INTERVENTIONS:
Procedure: Pleural drainage procedure with Seldinger procedure — Pleural drainage using Seldinger technique.
  Arms: Seldinger Technique
Procedure: Pleural drainage procedure with surgical-like technique — Pleural drainage using Surgical-like technique.
  Arms: Surgical-like Technique

SUMMARY:
This prospective randomized multicenter study is intended to investigate tolerance and effectiveness of thoracic drainage conducted by Seldinger technique with small drains, or by a surgical-like technique with large armed drains, in intensive care units patients.

DETAILED DESCRIPTION:
Drainage of pleural effusion and pneumothorax is a common feature in Resuscitation, Intensive Care Units (ICU) and Continuing Care Units (CCU). Although they are associated with a low incidence of complications (ranging from 0 to 8%), some of these can become fatal if they are associated with a visceral puncture (liver, spleen, lung parenchyma or heart by instance). It has been reported in the literature that complications were greater in case of drainage with large diameter drains set up by so-called "surgical-like" technique.

The choice of the type of chest tube is usually guided by the indication of drainage or the habits and / or experience of the practitioner. In the case of liquid pleural effusions, it may be preferable to use small diameter drains, whereas in the case of suspicious thick effusions such as empyema or blood, it may be preferable to use drainage drains of a larger diameter. However, results of retrospective analyzes seem to suggest the versatile and effective use of small-bore chest tubes in any of these indications without increasing complications' rates such as clogging.

However, no prospective randomized controlled trial (RCT) has studied this issue to date. Therefore, the investigators propose to perform a multicenter RCT in ICU and CCU patients requiring pleural drainage for any indication or underlying disease.

This prospective RCT is intended to investigate tolerance and effectiveness of thoracic drainage conducted by Seldinger technique with small drains, or by a surgical-like technique with large armed drains. Furthermore, they want to estimate the respective costs, identify the difficulties related to both strategies, recognize associated practices (ultrasound-guidance, implantation site, operator's competence), and finally point out the secondary determinants of tolerance and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Of-age patient (>18years)
* Patient admitted in ICU or CCU
* Patient requiring a pleural drainage, semi-urgent or planned
* Patient with a social security insurance

Exclusion Criteria:

* Patient under guardianship
* Severe or uncompensated bleeding disorders
* Thoracic trauma at the acute phase (<6 hours)
* Compressive pneumothorax requiring immediate and urgent needle exsufflation
* No thoracic drainage (whatever the technique used) performed previously during the same stay in ICU or CCU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Composite criteria of major and minor complications related to chest drainage | ICU discharge up to 6 months
  1. a composite criterion for major complications: organic lesions (spleen, liver, lung, artery, vessel ..., calculated frequency 0.2-1.4%) and post-drainage empyema or infection at the site level insertion rate (calculated frequency 0.2-1.4%) (non-inferiority hypothesis) and
  2. a composite criterion on the other complications (malposition of the drain (calculated frequency of 0.6-6.5%), clogging of the drain (calculated frequency of 8.1-5.2%) or drain drop (calculated frequency 1-21%) (hypothesis of superiority).

SECONDARY OUTCOMES:
Sedation and analgesia doses | Before, during, immediately after the procedure, every day until the removal of the chest tube, immediately after ICU discharge, Day 28 and Day 90
  Sedation and analgesia doses
Persistent residual pain: numerical pain scale | ICU discharge up to 6 months
  Evaluated by a numerical pain scale (VAS : 0 = No pain to 10 = Worst possible pain)
Evaluation of pain type | Before, during, immediately after the procedure, every day until the removal of the chest tube, immediately after ICU discharge, Day 28 and Day 90
  Type of pain neuropathic, nociceptive
Evaluation of Pain | Before, during, immediately after the procedure
  Evaluated by a numerical pain scale (if the patient is unable to communicate), or the BPS-NI (behavioral pain scale non-intubated, if the patient is non-intubated and unable to communicate, 3 to 12), or the BPS (behavorial pain scale, if the patient is intubated and unable to communicate, 0 to 12).
Procedural criteria | Immediately after the pleural drainage procedure
  Number of failures of the procedure
Procedural criteria | Immediately after the pleural drainage procedure
  Number of second operator necessary
Procedural criteria | Immediately after the pleural drainage procedure
  Number of drainage technique changes (cross-over)
Ultrasound use | Before, during and immediately after the pleural drainage procedure
  Rate of procedure use by care-providers
Ultrasound use | Before the pleural drainage procedure
  Volume to be drained according to published methods
Ultrasound use | Immediately after the pleural drainage procedure
  Assessment of pleural fluid type according to published methods
Ultrasound use | Immediately after the pleural drainage procedure
  Control of the position of the drain
General characteristics | Immediately after the pleural drainage procedure
  Type of Indication of drainage
General characteristics | Immediately after the pleural drainage procedure
  Diameter of drain used (millimeter)
General characteristics | Immediately after the pleural drainage procedure
  Diameter and brand of drain used
General characteristics | Immediately after the pleural drainage procedure
  Drainage duration
General characteristics | Immediately after the pleural drainage procedure
  Drain hold time in place
General characteristics | Immediately after the pleural drainage procedure
  Drain insertion site (safety triangle)
General characteristics | Immediately after the pleural drainage procedure
  Use or not of probabilistic antibioprophylaxis
General characteristics | Immediately after the pleural drainage procedure
  Number of differences between the result of the randomization and the doctor's choice in terms of drainage technique
Doctor performing drainage | Immediately after the pleural drainage procedure
  Characteristic's rate (senior or junior, prior experience with drainage technique)
General characteristics | Immediately after the pleural drainage procedure
  Rate of Off-hours drainage
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Infections at the insertion site or of pleural cavity during the ICU stay
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Post-drainage pneumothorax during the ICU stay
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Clogging of drain during the ICU stay
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Drain Malposition during the ICU stay
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Initiation of post-drainage mechanical ventilation if initially absent during the ICU stay
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Per- and post-procedure bleeding during the ICU stay during the ICU stay
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Intra- and post-drainage visceral lesions during the ICU stay
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Fall of the drain during the stay during the ICU stay
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Bad side or drainage site during the ICU stay
Complications' rates | During the pleural drainage procedure and ICU discharge up to 6 months
  Complications associated with drainages made on hold during the ICU stay
Patients outcomes | 6 months
  ICU mortality
Patients outcomes | 6 months
  Hospital mortality
Patients outcomes | Day 28
  ICU mortality
Patients outcomes | Day 28
  Hospital mortality
Patients outcomes | Day 28
  Days without mechanical ventilation
Patients outcomes | Day 90
  Days without mechanical ventilation
Patients outcomes | Day 90
  ICU mortality
Patients outcomes | Day 90
  Hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided